CLINICAL TRIAL: NCT00881738
Title: A Relative Bioavailability of Clarithromycin 250 mg Tablets Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Clarithromycin 250 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B013720
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Antibiotic
MeSH Terms: interventions — Clarithromycin

ARMS (2):
- 1 (Experimental): Clarithromycin 250 mg Tablets (Geneva, USA)
  Interventions: Drug: Clarithromycin 250 mg Tablets (Geneva, USA)
- 2 (Active Comparator): Biaxin 250 mg Tablets (Abbott Laboratories, Inc, USA)
  Interventions: Drug: Biaxin 250 mg Tablets (Abbott Laboratories, Inc, USA)

INTERVENTIONS:
Drug: Clarithromycin 250 mg Tablets (Geneva, USA)
  Arms: 1
Drug: Biaxin 250 mg Tablets (Abbott Laboratories, Inc, USA)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Clarithromycin 250 mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2002-06; Primary Completion 2002-06 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services